CLINICAL TRIAL: NCT01281527
Title: A 6-month, Open Label, Prospective, Multicenter, International, Exploratory Study of a Transition to Flexibly Dosed Paliperidone Palmitate in Patients With Schizophrenia Previously Unsuccessfully Treated With Oral or Long-acting Injectable Antipsychotics
Brief Title: Paliperidone Palmitate Flexible Dosing in Schizophrenia
Acronym: PALMFlexS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017215; R092670SCH3010 (Other: Janssen-Cilag International)
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Schizophrenia
Keywords: Paliperidone palmitate; Schizophrenia; Intramuscular injection
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paliperidone Palmitate (Experimental): Paliperidone Palmitate 50 - 150 mg eq. every 30 days for 6 months during the core phase and for 12 months during an optional extension phase after the last patient has completed the 6-month core treatment phase or until product will be available on market (whichever comes first)
  Interventions: Drug: Paliperidone Palmitate

INTERVENTIONS:
Drug: Paliperidone Palmitate — 50 - 150 mg eq. every 30 days

SUMMARY:
This study explores the tolerability, safety and efficacy (i.e. how well the drug works) of flexibly dosed paliperidone palmitate in the treatment of schizophrenia in patients previously unsuccessfully treated with other oral or long-acting injectable (LAI) (i.e. with a long duration of action) antipsychotics.

DETAILED DESCRIPTION:
This study explores the tolerability, safety and treatment response of flexibly dosed paliperidone palmitate in approximately 1,000 patients with schizophrenia previously unsuccessfully treated with an oral or LAI antipsychotic medication. Non-acute and acute patients will be involved in the study. This study consists of a screening phase, a 6-month core treatment phase, and an optional extension phase. A transition period of preferably a maximum of 4 weeks will be allowed for the previous oral antipsychotic. When switching patients from previous LAI antipsychotics, paliperidone palmitate will be initiated in place of the next scheduled injection. Patients without source documentation of previous risperidone or paliperidone exposure must undergo oral tolerability testing with paliperidone ER (3 mg/day) for the 2 days prior to Baseline Visit. Patients who successfully complete the 6-month core treatment phase and would like to continue treatment with paliperidone palmitate may be enrolled in an optional extension phase until paliperidone palmitate is available in their respective country or until a maximum duration of 12 months after the last subject has completed the 6-month core treatment phase, whichever comes first. Patients will receive, without cost, paliperidone palmitate. Patients entering this optional extension phase, will receive once monthly injections with paliperidone palmitate. The recommended maintenance dose for these monthly injections is 75 mg eq. once monthly but flexible dosing in the range of 50 to 150 mg eq. once monthly will be allowed. The doctor may flexibly increase or decrease the dose preferably by one dosing level (within the range of 50 to 150 mg eq.) according to patients' clinical needs. During the extension phase, two types of visits can be distinguished: 'assessment visits' and 'treatment-only visits'. At each assessment visit (once every 3 months +/- 7 days), patients will receive their injection and will be questioned about adverse events (AEs). Body weight will also be assessed. Paliperidone palmitate will be given once monthly by injection in either the upper arm or buttocks muscle, but start every time with upper arm application. The recommended maintenance dose for these monthly injections is 75 mg eq., range could be between 50 to 150 mg eq.

ELIGIBILITY:
Inclusion Criteria:

Meet the DSM-IV criteria for schizophrenia Currently non-acute, i.e., on the same antipsychotic medication used for the treatment of schizophrenia given in an adequate dose and a CGI-S change <= 1 in the past 4 weeks before enrollment Patient has been given an adequate dose of either an appropriate oral antipsychotic, or a protocol-defined LAI antipsychotic for an adequate period of time prior to enrollment, but current treatment is considered unsuccessful OR Patients with acute symptoms of schizophrenia, previously treated with an oral antipsychotic, having a baseline total Positive and Negative Syndrome Scale (PANSS) score >= 80 and a baseline CGI-S score >= 4 Women must be postmenopausal for at least 1 year, surgically sterile, abstinent (at the discretion of the investigator/per local regulations), or if sexually active, be practicing a highly effective method of birth control as local regulations permit, and before entry, must agree to continue to use the same method of contraception throughout the study Is cooperative and reliable, and agrees to receive regular injections and complete all aspects of the protocol Men must agree to use a double barrier method of birth control and to not donate sperm during the study and for 3 months after receiving the last dose of study drug.

Exclusion Criteria:

The patient's psychiatric diagnosis is due to direct pharmacological effects of a substance (e.g., a drug of abuse or medication) or a general medical condition (e.g., clinically notable hypothyroidism) First antipsychotic treatment ever, i.e., patient has never been treated with antipsychotics before and antipsychotic treatment given in this study will be the first antipsychotic treatment that the patient will have ever received On clozapine during the last 3 months Patients who remain at imminent risk of suicide even after clinical intervention Serious unstable medical condition, including recent and present clinically relevant laboratory abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1044 (Actual)
Dates: Start 2010-11; Primary Completion 2012-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Improved efficacy for non-acute patients transitioned due to lack of efficacy, as measured by the total PANSS score at endpoint versus baseline. | Baseline to 6 months or early discontinuation
Improved efficacy for acute patients, as measured by the total PANSS score at endpoint versus baseline. | Baseline to 6 months or early discontinuation
Maintained efficacy for non-acute patients transitioned for other reasons based on PANSS score at endpoint versus baseline. | Baseline to 6 months or early discontinuation

SECONDARY OUTCOMES:
Change from baseline in Clinical Global Impression-Severity Scale [CGI-S] | Baseline, week 1, month 1, 2, 3 and 6
Change from baseline in personal and social functioning (Personal and Social Performance Scale [PSP]) | Baseline, week 1, month 1, 2, 3 and 6
Change from baseline in Health status (Self-reported health status questionnaire [SF-36]) | Baseline, month 3 and 6
Change from baseline in Measure of Health Outcome (EQ-5D) | Baseline, month 3 and 6
Change from baseline in Patient well-being (Subjective Well-Being under Neuroleptics Scale [SWN-S]); | Baseline, month 3 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (127):
- Salzburg, Austria
- Belgium (9):
  - Brussels
  - Dave
  - Diest
  - Kruishoutem
  - Liège
  - Melle
  - Roeselare
  - Sint-Denijs-Westrem
  - Tournai
- Croatia (2):
  - Rijeka
  - Zagreb
- Denmark (3):
  - Aalborg
  - København V
  - Randers
- Tallinn, Estonia
- France (15):
  - Bar-le-Duc
  - Bron
  - Clermont-Ferrand
  - Dax
  - Dijon
  - Dole
  - Lille
  - Limoges
  - Montpellier
  - Nîmes
  - Paris
  - Saint-Nazaire
  - Saint-Priest-en-Jarez
  - Strasbourg
  - Villejuif
- Germany (18):
  - Bad Saarow
  - Berlin
  - Bielefeld
  - Bochum
  - Butzbach
  - Dresden
  - Gelsenkirchen
  - Greifswald
  - Hamburg
  - Heidelberg
  - Königsbrück
  - Mittweida
  - Oranienburg
  - Regensburg
  - Stralsund
  - Ulm
  - Westerstede
  - Würzburg
- Greece (5):
  - Arta
  - Athens
  - Katerini
  - Thessaloniki
  - Thessalonikis
- Hungary (3):
  - Budapest
  - Debrecen
  - Pécs
- Israel (3):
  - Pardesiyya
  - Ramat Gan
  - Tirat Hacarmel
- Latvia (6):
  - Daugavpils
  - Jelgava
  - Liepāja
  - Riga
  - Sigulda
  - Strenči
- Lithuania (2):
  - Panevezys
  - Vilnius
- Groningen, Netherlands
- Portugal (6):
  - Almada
  - Angra do Heroísmo
  - Castelo Viegas
  - Coimbra
  - Lisbon
  - Porto
- Spain (15):
  - Alcorcón
  - Alicante
  - Barcelona
  - Burgos
  - Coslada
  - Elche
  - Madrid
  - Málaga
  - Palma de Mallorca
  - Sant Boi de Llobregat
  - Sant Joan d'Alacant
  - Santa Coloma de Gramenet
  - Vigo
  - Zamora
  - Zaragoza
- Sweden (6):
  - Gothenburg
  - Lidingö
  - Malmo
  - Mölndal
  - Spånga
  - Upplands Vasby
- Switzerland (2):
  - Solothurn
  - Zurich
- Turkey (Türkiye) (6):
  - Ankara
  - Diyarbakır
  - Gaziantep
  - Istanbul
  - Izmir
  - Trabzon
- Ukraine (14):
  - Dnipro
  - Donetsk
  - Hlevakha
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Lviv
  - Odesa
  - Poltava
  - Simferopol
  - Smila
  - Ternopil
  - Uzhhorod
  - Yevpatoria
- United Kingdom (9):
  - Barnet
  - Birmingham
  - Cambridge
  - Coventry
  - Darlington
  - Lincoln
  - London
  - Prescott
  - Stoke-on-Trent

REFERENCES:
- [Derived] Schreiner A, Bergmans P, Cherubin P, Keim S, Rancans E, Bez Y, Parellada E, Carpiniello B, Vidailhet P, Hargarter L. A prospective flexible-dose study of paliperidone palmitate in nonacute but symptomatic patients with schizophrenia previously unsuccessfully treated with oral antipsychotic agents. Clin Ther. 2014 Oct 1;36(10):1372-88.e1. doi: 10.1016/j.clinthera.2014.08.014. Epub 2014 Oct 23. PMID 25444566
- See also: A 6-Month, Open-Label, Prospective, Multicenter, International, Exploratory Study of a Transition to Flexibly-Dosed Paliperidone Palmitate in Patients with Schizophrenia Previously Unsuccessfully Treated with Oral or Long-Acting Injectable Antipsychotics — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=229&filename=CR017215_CSR.pdf